CLINICAL TRIAL: NCT00382772
Title: Study to Evaluate Clinical Consistency of the Liquid Formulation of GSK Biologicals' HRV Vaccine and to Evaluate Liquid Formulation Compared to Lyophilised Formulation of the HRV Vaccine Administered as a Two-dose Primary Vaccination.
Brief Title: A Study in Infants to Test Two Preparations (Freeze-dried or Liquid) of the Rotavirus Vaccine (HRV Vaccine).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107876
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Rotavirus
Keywords: HRV vaccine; Diarrhoea; Rotavirus
MeSH Terms: conditions — Rotavirus Infections; Diarrhea

INTERVENTIONS:
Biological: 2-dose oral live attenuated G1P[8] human rotavirus vaccine

SUMMARY:
The aim of this this study is to evaluate the lot-to-lot consistency of the liquid formulation of GSK Biologicals' HRV vaccine and to evaluate the liquid formulation compared to the lyophilised formulation of GSK Biologicals' HRV vaccine when administered concomitantly with a combination childhood vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants birth weigh >2000 g, 11 -17 weeks old at Dose 1 with written informed consent.

Exclusion Criteria:

* Allergic reaction to vaccine components; clinically significant history of chronic GI disease (uncorrected GI congenital malformation) or other serious medical condition per investigator, received vaccines or treatment prohibited by the protocol; immunocompromised.

Ages: 11 Weeks to 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Demonstrate lot-to-lot consistency of HRV vaccine liquid formulation and non-inferiority of liquid formulation versus the lyophilised formulation of the HRV vaccine.

SECONDARY OUTCOMES:
Assess lot-to-lot consistency in terms of reactogenicity and assess safety of HRV vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Finland (10):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Vesikari T, Karvonen A, Bouckenooghe A, Suryakiran PV, Smolenov I, Han HH. Immunogenicity, reactogenicity and safety of the human rotavirus vaccine RIX4414 oral suspension (liquid formulation) in Finnish infants. Vaccine. 2011 Mar 3;29(11):2079-84. doi: 10.1016/j.vaccine.2011.01.004. Epub 2011 Jan 14. PMID 21238572
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 107876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107876 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register